CLINICAL TRIAL: NCT06642974
Title: Development, Validation and Testing of an Education Program for Identification of Learning Disabilities Among School Children by Primary School Teachers in Qatar
Acronym: LD - Learning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Ramya Munuswamy, Nurse Educator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MRC-01-23-170
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Learning Disabilities, Child
Keywords: Learning Disabilities, children
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: experimental and control group, experimental group will receive formal education control group will receive informative pamphlets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental - Education module on Learning disabuilities (Experimental): A total of 67 samples will receive the education module delivery on early identification of learning disabilities
  Interventions: Other: Education module on learning disabilities
- Control (Other): A total of 67 samples will receive education pamphlets on early identification of learning disability
  Interventions: Other: pamphlet on learning disability

INTERVENTIONS:
Other: Education module on learning disabilities — Data will be collected for a period of one -year. samples will be equally distributed among experimental and control group. Socio -demographic data and knowledge and attitude of primary school teachers on learning disability will be assessed by interview method using questionnaire. Control group will receive general information on children with learning disabilities while experimental group will receive education training program. After 15 days again education program will be repeated as a reinforcement. Pre and posttest will be conducted for both the groups at one-month interval. Required data will be collected for one-year period by interview method using questionnaire. Competency assessment will be done by using checklist on identification of learning disabilities Teachers' competency for experimental group then the competency will be verified by education counselor . As a follow up of the research study, after one-month interval no of referral by each teacher will be collected to m
  Arms: Experimental - Education module on Learning disabuilities
Other: pamphlet on learning disability — Education pamphlets will be provided to total of 67 samples
  Arms: Control

SUMMARY:
Aim The aim of this study to develop, validate and test an education program for identification of learning disabilities among school children by Primary school teachers in Qatar Objectives

1. To develop and validate an education program on identification of learning disabilities of children by primary school teachers
2. To evaluate the effectiveness of an education program regarding identification of learning disabilities of children.

DETAILED DESCRIPTION:
Education is one of the essential aspects of the growth of children. At the right time, each child must get the right education. The aim of education is to educate the child in a way that promotes the interest and needs of the child. Each child has unique learning styles. Learning is any ongoing shift in action that happens because of practice and experience. As this is indicated in Qatar's national policy every child should be provided with education to help it reach its full potential.

Learning disability (LD) is a worldwide problem today. According to American Psychiatric Association (2018) an estimated 5 to 15 percent school age children struggle with a LD.As stated by fifth edition of Diagnostic and Statistical manual of Mental Disorders (DSM-V-R,2013), learning disabilities refer to the conditions when academic skills are greatly below the average range of expected scores based on the chronological age (e.g. at least 1.5 SD below the population mean score for age). The difference between intelligence and academic achievement scores in standardized reading, mathematical tests, and written expressions is basically lower than the chronological age, intellectual, and educational level. The learning problems significantly interfere with academic achievement or activities of daily living that require reading, mathematical or writing skills". Common learning disabilities dyslexia, dyscalculia, dysgraphia, auditory and visual processing disorder, and nonverbal learning disabilities.

Teachers plays an important role in all educational system. Teacher is an originator who creates and forms children's physical, intellectual, and moral capacity, which gives teachers tremendous obligation to train themselves to recognize children at regular school with learning disabilities Each classroom has one or two children with learning disabilities at a regular school. The ability of teachers to assess learning disabilities in normal schools is a key factor. This needs teachers to undergo an additional training program to recognize primary-level children with LD.

Need for the study Learning disability is the largest disability among school going children with prevalence rate between 3% and 12% in elementary school students. Most of the students attend regular school due to misdiagnosis of intellectual disability. Those who attend regular schools face many challenges in educational progress, even they have school failure. LD is the main contributing factor in which 37.9% for school failure in Qatar. This results in low self -esteem, difficulty in learning can continue in adolescent age and later children stop studying to learn eventually drop out of school.

One of the most important strategies for an early detection of these abnormalities is to be referring them by primary school teachers to an educational counselor, including speech therapists, for an adequate and thorough assessment and the final diagnosis of childhood LD. This allows teachers to be mindful of LD signs and symptoms and to perform initial student screening. Otherwise, assessment and diagnosis can be delayed or lead to adverse outcomes. Therefore, awareness and attitude of primary school teacher about LD are very important.

As Qatar's expat > 85% (What makes an effective teacher, ex. summary, Katherine McKnight), population has grown exponentially. so, too, has the number of private schools. There are schools established for almost every nationality: American, British Canadian, French, German, Indian, Filipino, and Lebanese. However, the rise in the number of private schools has not contributed to a proportionate increase in the standard of private schools. This is due to teachers leaving the job in between the academic year on varied reasons. (Education in Doha, Qatar: an overview, The Good School Guide newsletter) As this results in, the same teachers to track students on the entire grade will be missed. So, there are chances for in identifying LD in primary school level will be challenging.

It has been noted that many schools in Qatar employs a large number of teachers from other countries, it would be beneficial to understand the level of knowledge of teachers from different countries who might have different amount of training and experience. Also, it gives baseline data to education legislators to plan additional educational activities to improve primary school teachers' knowledge and practice on identifying children with LD.

Ministry of Education and Higher Education and Supreme Education Council, Qatar is committed to inclusive integration in education where possible. Some 80% of independent schools have introduced additional educational needs facilities and staffs. Additional to that many workshops and in-service programs are held for teachers in order to educate the children with special needs including learning disabilities in private schools, such program help with identifying signs and symptoms in a timely manner. However, it requires the institute, or government should arrange appropriate training or structured teachers program covering aspects of these dimensions about concept, diagnosing, and identifying special students with learning problems. Identifying and assessing primary school teachers' knowledge level is very important aspect in before developing an educational program, thus it gives an opportunity to design the educational program according to teacher's knowledge level. Developing and implementing education module is an important strategy to utilize teachers as effective contributors towards child health services. This emphasis there is huge requirement to develop an educational program for primary school teachers to identify children with LD in regular school.

Teachers' previous knowledge and basic education program provides some knowledge about learning disability, such knowledge was grossly insufficient for its practical application in the classroom. This indicates that some teachers were not adequately equipped to identify and remediate learning disability in the classroom. Hence this identifies competency assessment is an essential element to be assessed along with education program. Competency assessment increases the level of competency of professional teachers to recognize alleged cases of learning disabilities. learning package improves the competency of primary school teachers regarding learning disabilities and understanding of teachers' competency includes definition of teachers' competency, teachers' role in identifying children at risk of LD. While discussing the importance of identifying LD at primary school children by teachers' until now, no such research has been conducted in Qatar upon the level of knowledge, attitude and competence among primary school teachers in identifying children with LD. Therefore, the present study is planned to develop, validate and test an education program and screening tool for identification of learning disabilities among school children by Primary school teachers in Qatar

The purpose of the study is to develop and validate education program for primary school teachers to identify LD, this focus group discussion will guide to structure the questionnaire to assess the teacher's knowledge level and develop and validate education module on LD

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

The study will include:

* Teachers who are teaching in private schools in state of Qatar
* Teachers who are teaching Indian curriculum
* Teachers who are teaching subjects such as English, mathematics, environmental science, and science
* Teachers who can speak and write English.

Exclusion Criteria:

* Teachers who are not willing to participate in the study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary school teachers' knowledge level will increase | 4 weeks
  At the end of the Research study,
  * A validated and tested education program will be available for use by primary school teachers
  * Teacher's Knowledge on identifying LD will increase
  * Teacher's Competency level in identifying LD will improve
  * There will be increased number of referrals and early diagnosis of LD

IPD SHARING:
Plan to Share IPD: No
Data will be kept with principle investigator ; no unauthorized person will have access to it at any stage of the study. Special precautions will be followed to maintain the anonymity of the participants.
  Data will be stored in HMC and personal computer with passcode lock